CLINICAL TRIAL: NCT06012422
Title: Sarcopenia Screening in Elderly Individuals Living in Kirikkale Province
Brief Title: Sarcopenia Screening in Elderly Individuals
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kırıkkale University (Other)
Responsible Party: Principal Investigator, Seyma Akdagli, Master of Science Student, Kırıkkale University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: KU-FTR-SA-01
Record Dates: First submitted 2023-08-20; First posted 2023-08-25 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Sarcopenia
Keywords: rehabilitation; physical inactivity; fragility
MeSH Terms: conditions — Sarcopenia; Sedentary Behavior

STUDY DESIGN:
Intervention Model Description: There is no randomization in our study, all elderly individuals who meet the inclusion and exclusion criteria will be evaluated.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Individuals aged 65 and over who were screened for sarcopenia (Other): Persons aged 65 and over will be evaluated only once and the assessment will be made through a face-to-face interview.
  Interventions: Other: evaluation group

INTERVENTIONS:
Other: evaluation group — Elderly individuals will be evaluated once, by face-to-face interview method.

SUMMARY:
In this study, it is aimed to evaluate parameters such as sarcopenia screening, muscle mass measurement, loss of strength that may develop due to sarcopenia, loss of balance and related fall, decrease in functionality, fragility and decreased physical activity in individuals aged 65 years and older in Kırıkkale city center.

DETAILED DESCRIPTION:
Although aging occurs in all periods in the human body, physical, mental and physical aging becomes visible as you get older. This situation is caused by physiological aging, environmental factors, existing chronic diseases and related symptoms. Today, increasing life expectancy and aging population must be taken into account. Since the age-related symptoms of elderly individuals are compatible with the consequences of aging, they can be ignored as a natural process, and therefore its progression cannot be prevented. With our project, it is aimed that screening for sarcopenia will be an exemplary study throughout Turkey and this type of screening will be widespread. In addition, it is aimed to divide elderly individuals into groups as presarcopenia, sarcopenia and severe sarcopenia, and to provide necessary guidance, protective and prevention approaches, strengthening and exercise training.

Demographic data of elderly individuals (age, gender, height, weight, BMI (Body mass index will be obtained by dividing body weight (kg), height (m) squared) occupation, etc.), chronic diseases (hypertension, diabetes, chronic obstructive pulmonary disease) (COPD), rheumatic diseases), drugs used, smoking, alcohol habits, and assistive device use, and the 'Clinical Vulnerability Scale' to evaluate the cognitive status of individuals through the 'Mini Nutritional Assessment form (MNA)'. 'Standardized Mini-Mental Test' to assess balance and walking, 'Tinetti balance and walking test' to evaluate balance and walking, 'Falling Risk Self-Assessment Scale' to assess falls, 'Functional Independence and Challenge Scale' to measure functional independence in activities of daily living. 'Short Physical Performance Test' (KFPT), Sarcopenia screening test (SA) to assess physical fitness RC-F), it is planned to use the Physical Activity Scale for the Elderly (PASE) to evaluate the level of physical activity, to use hand dynamometer, to evaluate muscle strength, and to measure the muscle mass of individuals with an inbody bioimpedance device.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 65 and over
* Their willingness to participate in the study
* A score of 24 or higher on the Mini Mental State Test (MMDT)

Exclusion Criteria:

* Individuals under the age of 65
* Individuals who cannot communicate well
* Elderly individuals who cannot walk independently, have any orthopedic or neurological problems
* Individuals who do not want to participate in the study
* Individuals not eligible for bioimpedance analysis (pregnant individuals with pacemakers).

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 843 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2023-10-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Bioimpedance Analysis | day 1
  used to measure muscle mass in epidemiological studies.A muscle mass index of less than 5.5 in women and less than 7 in men is associated with the risk of sarcopenia.

SECONDARY OUTCOMES:
Muscle Strength Evaluation | day 1
  Handgrip strength is more commonly used, and low handgrip strength correlates better with impaired mobility and undesirable clinical outcomes than low muscle mass. In practice, a linear relationship was also found between basal handshake strength and dependence on activities of daily living. Therefore, hand grip strength measurement is a good and simple method to evaluate muscle strength.
Short Physical Performance Test | day 1
  The test measures parameters such as balance, sitting and standing from a chair and walking speed.All three physical performance measures (walking speed, balance, getting up from a chair) are scored between 0-4 according to the duration of the activity, the scores of the three tests are summed to give a total score between 0 (poor) and 12 (very good).
SARC-F | day 1
  Used for rapid diagnosis of sarcopenia.In the SARC-F questionnaire, information such as strength, walking without support, getting up from a chair/stool, climbing stairs and the number of falls in the last year are questioned (66). According to the EWGSOP2 guideline, a score of 4 or higher on the SARC-F questionnaire is considered significant in terms of sarcopenia.
Mini Nutritional Assessment | day 1
  The long MNA contains 18 items collected in 4 chapters. These four parts; anthropometric assessment (BMI, weight, arm and calf circumferences); overall assessment (lifestyle, medication, mobility, depression and dementia symptoms); short nutritional assessment (number of meals, food and fluid intake, autonomy in nutrition) and subjective assessment (self-perception of health and nutrition)
Physical Activity Scale for the Elderly | day 1
  The questionnaire evaluates the physical activities of the bereaved individuals in the last week and includes the components of leisure time, housework and work-related physical activity. walking activity outside the home; mild, moderate and vigorous sports and recreational activities; Participation in leisure time activities, including muscle strengthening exercises, was recorded as never, rarely (1-2 days / week), sometimes (3-4 days / week), and often (5-7 days / week), while the duration of the activities was: 1 It is classified as less than 1 hour, 1-2 hours, 2-4 hours and more than 4 hours.
Tinetti balance and walking test | day 1
  assesses balance and walking.In the test, the walking score is a maximum of 12 points, the balance score is a maximum of 16 points, and a total of 28 points. Those who score twenty-six and below are considered to have a problem. Studies have shown that the risk of falling increases as the score decreases.
Fall Risk Self-Assessment Scale | day 1
  It is a scale that assesses the risk of falling in the elderly. It consists of 13 items assessing the risk of falling in the elderly. The answers are yes (1 point) and no (0 points), and individuals who get 4 points or more from the score are classified as having a high risk of falling.
Anthropometric Measurements | day 1
  Anthropometric measurements of middle arm muscle circumference and calf circumference have been shown to predict functionality, general health status, nutritional adequacy, and survival in the elderly.
  It has been reported that calf circumference of 31 cm or less, arm circumference of 23 cm or less in women, and 24 cm or less in men are associated with sarcopenia.